CLINICAL TRIAL: NCT01681147
Title: Barriers to Adherence to Recommended Follow-up in Women With a History of Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS 2012-16
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes; postpartum; nutrition; exercise
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care (No Intervention): Standard postpartum care after a pregnancy with gestational diabetes
- Standard Care+Education Classes (Experimental): Standard postpartum care after a pregnancy with gestational diabetes
  2 online nutrition and exercise education classes
  Interventions: Behavioral: 2 online nutrition and exercise education classes
- Standard Care+Education Classes+Glucose Monitoring (Experimental): Standard postpartum care after a pregnancy with gestational diabetes
  2 online nutrition and exercise education classes
  Self monitoring of blood glucose levels
  Interventions: Behavioral: 2 online nutrition and exercise education classes; Behavioral: Self monitoring of blood glucose levels

INTERVENTIONS:
Behavioral: 2 online nutrition and exercise education classes — Two online nutrition and physical activity classes will accessed from a computer, android phone or a tablet. Each class is estimated to last about 1.5- 2 hours and will be accessed 6 weeks-3 months and 9 months
  Arms: Standard Care+Education Classes; Standard Care+Education Classes+Glucose Monitoring
Behavioral: Self monitoring of blood glucose levels — Self monitoring of blood glucose levels four times a day for four consecutive days once a month from 6 weeks-3 months through 9 months post partum
  Arms: Standard Care+Education Classes+Glucose Monitoring

SUMMARY:
The purpose of this study is to find out whether women who have had gestational diabetes mellitus (GDM) will make healthier lifestyle choices, achieve weight goals, and complete postpartum care assessments after receiving two online classes on healthy nutrition and exercise classes at 6 weeks - 3 months and at 9 months postpartum.

DETAILED DESCRIPTION:
For this pilot study, we propose to conduct a 3-grouped randomized controlled trial to evaluate whether a 1 ½ to 2 hour on-line nutrition and physical activity intervention +/- block testing of blood glucoses fasting and 2 hours after each meal for 4 days/month from starting at 3 months postpartum and concluding at 9 months postpartum will: 1) improve adherence to the receipt of diabetes screening at 12 months postpartum through the recommended 75 gram 2 hour oral glucose tolerance test (OGTT) or fasting blood glucose test, 2) lower glucose values on the 75 gram 2 hour oral glucose tolerance test or fasting blood glucose test and 3) improve attainment of weight loss targets among women with a recent history of GDM.

Patients will participate in an online nutrition and physical activity class from 6 weeks to 3 months and 9 months for women assigned to both groups 2 and 3. For those women assigned to group 3, they will also do block testing using an assigned blood glucose meter and test strips 4 times a day for 4 consecutive days each month, starting at 3 months and ending at 9 months. Women will have the option of submitting meter blood glucose data via e-mailed logs or downloading directly to the clinic using Diasend software. Once downloaded, the Diasend software will create a PDF document with all recorded blood glucose values.

For purposes of this study, we will obtain a Diasend account specific to this study, which will allow women to download blood glucose information with an anonymous unique identifier that can be accessed by the study's Principal Investigator and the Collaborative Institutional Training Initiative (CITI)-certified, International Review Board (IRB)-approved research assistant. Upon accessing the PDF document with the blood glucose meter information, both the PI and the Research Assistant can link blood glucose data with questionnaire and other health information collected in this study through the unique identifiers.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Diabetes
* Age between 21 and 45 years
* Preconception BMI 19-40
* Seen for at least 2 visits in the Diabetes in Pregnancy Program during their pregnancy
* Singleton pregnancy

Exclusion Criteria:

* Preexisting diabetes or diabetes diagnosed at the 6 week 75 gram 2 hour OGTT
* BMI >40
* Multiple gestation (i.e., twins, triplets, etc.)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Brown, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Originally, the number of participants in each of the arms was supposed to be 10 participants per arm. However, due to assignment error, Group 2 only received 8 participants and Group 3 received an additional 2.
Groups:
- Standard Care+Education Classes: Standard postpartum care after a pregnancy with gestational diabetes
  2 online nutrition and exercise education classes
  2 online nutrition and exercise education classes: Two online nutrition and physical activity classes will accessed from a computer, android phone or a tablet. Each class is estimated to last about 1.5- 2 hours and will be accessed 6 weeks-3 months and 9 months
- Standard Care+Education Classes+Glucose Monitoring: Standard postpartum care after a pregnancy with gestational diabetes
  2 online nutrition and exercise education classes
  Self monitoring of blood glucose levels
  2 online nutrition and exercise education classes: Two online nutrition and physical activity classes will accessed from a computer, android phone or a tablet. Each class is estimated to last about 1.5- 2 hours and will be accessed 6 weeks-3 months and 9 months
  Self monitoring of blood glucose levels: Self monitoring of blood glucose levels four times a day for four consecutive days once a month from 6 weeks-3 months through 9 months post partum
Period: Overall Study
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Started | 10 | 8 | 12
Baseline | 9 | 7 | 10
3 Months | 8 | 5 | 8
6 Months | 7 | 6 | 7
9 Months | 7 | 5 | 6
12 Months | 5 | 4 | 5
Completed | 0 | 0 | 1
Not Completed | 10 | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring | Total
Number analyzed (Participants) | 10 | 8 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 12 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.3 [33.1 to 39.4] | 35.3 [34.2 to 38.9] | 34.6 [30.9 to 37.2] | 35.1 [32.6 to 37.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 12 | 30
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 6 | 9 | 24
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 2 | 0 | 2
  White | 5 | 1 | 8 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Women with a History of Gestational Diabetes [Count of Participants; unit: Participants] | 10 | 8 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: 1. Postpartum weight loss (target 7% less than the pre-pregnancy weight for overweight/obese women and back to pre-pregnancy weight for normal BMI women). This will be based on medical record information on pre-pregnancy weight and self-reported or health-care provider reported weight at 12 months.
Time Frame: 1 year postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Number analyzed (Participants) | 10 | 8 | 12
Participants | 0 | 0 | 2

2. Primary Outcome: Postpartum Diabetes Screening at One Year
Description: 1. Adherence to diabetes screening using the 75 gram 2 hour oral glucose tolerance test (OGTT) or fasting blood glucose at 12 months (+/- 3 months).
  2. Lab results from the fasting glucose test or results from a 75 gram 2 hour OGTT at 12 months among women who choose to take the diabetes screening test.
Time Frame: 1 year postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Number analyzed (Participants) | 10 | 8 | 12
Participants | 0 | 1 | 1

3. Primary Outcome: Barriers Associated With Poorer Adherence to Diabetes Screening Guidelines and Weight Loss Goals
Description: 2. Determine to what extent barriers to health impact adherence rates to post partum screening and weight loss targets through a web-based questionnaire collected on the 6 weeks to 3 months, 6, 9, and 12 month questionnaires. These questionnaires will assess whether: lack of self care, perception of high infant care giving needs, fear of diabetes diagnosis and postpartum depressive symptoms, difficulty accessing medical care, dissatisfaction with medical care or primary care physician not recommending screening are associated with poorer adherence to diabetes screening guidelines and weight loss goals.
Time Frame: Assessed at 6 weeks to 3 months, 6 months, 9 months, and 12 months, 6 months reported
Population: Lack of Self-Care, Infant Care: 1) Not at all 2) Seldom 3) Sometimes 4) Frequently 5) Always.
  Fear of Diabetes Diagnosis & PP Depression 1) Most of the time 2) Some of the time 3) Not very often 4) Not at all.
  Difficulty Accessing Medical Care, Dissatisfaction w/ Medical Care: 1) strongly disagree 2) disagree 3) Neutral 4) Agree 5) Strongly Agree
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Number analyzed (Participants) | 7 | 6 | 7
score on a scale
  Lack of Self-Care | 2.08 (0.61) | 2.20 (0.86) | 2.52 (0.57)
  Perception of High Infant Care Giving Needs | 1.60 (0.33) | 1.57 (0.50) | 1.97 (0.49)
  Fear of Diabetes Diagnosis & PP Depression | 2.99 (1.09) | 2.93 (0.97) | 2.83 (0.87)
  Difficulty of Accessing Medical Care | 3.3 (0.45) | 3.8 (0.84) | 3.3 (0.67)
  Dissatisfaction with Medical Care | 2.96 (0.89) | 3.08 (089) | 3.0 (1.08)

4. Secondary Outcome: Dietary Pattern Assessment of Women With Gestational Diabetes Postpartum
Description: Determine to what extent types of food products and amount of exercise frequented by women with gestational diabetes postpartum impacted adherence rates to weight loss targets through a web-based questionnaire collected at the 3 month, 6 month and 9 month follow-up. These questionnaires will assess whether eating patterns associated with poorer adherence to diabetes screening guidelines and weight loss goals.
Time Frame: 3 months, 6 months, 9 months, all reported
Population: Scale was ranked as follows: 1 = Never/Less than once a week; 2 = Once per week; 3 = 2 to 4 times per week; 4 = Nearly daily or daily; 5 = Twice or more per day Patients were asked to rank how often they ate certain types of foods (i.e. starches, vegetables, etc.). Individual questions were categorized into healthy vs. unhealthy neutral foods.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Number analyzed (Participants) | 10 | 8 | 12
score on a scale
  Frequency of Healthy Food (3 month): number analyzed (Participants) | 8 | 5 | 8
  Frequency of Healthy Food (3 month) | 2.46 (0.79) | 2.77 (0.92) | 2.4 (0.89)
  Frequency of Unhealthy Food (3 month): number analyzed (Participants) | 8 | 5 | 8
  Frequency of Unhealthy Food (3 month) | 1.57 (0.71) | 1.53 (0.73) | 1.69 (0.66)
  Frequency of Neutral Food (3 month): number analyzed (Participants) | 8 | 5 | 8
  Frequency of Neutral Food (3 month) | 1.94 (0.43) | 1.81 (0.70) | 1.75 (0.96)
  Frequency of Healthy Food (6 month): number analyzed (Participants) | 7 | 5 | 7
  Frequency of Healthy Food (6 month) | 2.52 (0.94) | 2.54 (0.83) | 2.46 (0.96)
  Frequency of Unhealthy Food (6 month): number analyzed (Participants) | 7 | 5 | 7
  Frequency of Unhealthy Food (6 month) | 1.53 (0.66) | 1.67 (0.71) | 1.70 (0.75)
  Frequency of Neutral Food (6 month): number analyzed (Participants) | 7 | 5 | 7
  Frequency of Neutral Food (6 month) | 1.89 (1.02) | 1.85 (0.72) | 2.11 (0.99)
  Frequency of Healthy Food (9 month): number analyzed (Participants) | 7 | 5 | 6
  Frequency of Healthy Food (9 month) | 2.56 (0.92) | 2.73 (0.80) | 2.58 (0.97)
  Frequency of Unhealthy Food (9 month): number analyzed (Participants) | 7 | 5 | 6
  Frequency of Unhealthy Food (9 month) | 1.52 (0.72) | 1.5 (0.51) | 1.68 (0.71)
  Frequency of Neutral Food (9 month): number analyzed (Participants) | 7 | 5 | 6
  Frequency of Neutral Food (9 month) | 1.89 (0.98) | 1.91 (0.93) | 2.04 (0.87)

5. Secondary Outcome: Food Frequency Questionnaire
Description: The table shows the percent of women eating each food daily or nearly daily.
Time Frame: 3 months, 6 months, 9 months, all reported
Population: The "Overall Number of Participants Analyzed" defines the number of participants enrolled in the study.
  The Number in the Rows indicates the number of participants that completed the follow-up surveys required for participation in the study.
Measure: Number; unit: % women eating food daily or near daily
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Number analyzed (Participants) | 10 | 8 | 12
% women eating food daily or near daily
  Leafy Greens (3 months): number analyzed (Participants) | 8 | 5 | 8
  Leafy Greens (3 months) | 87.5 | 20.0 | 50.0
  Leafy Greens (6 months): number analyzed (Participants) | 7 | 5 | 7
  Leafy Greens (6 months) | 57.1 | 60.0 | 42.9
  Leafy Greens (9 months): number analyzed (Participants) | 7 | 5 | 6
  Leafy Greens (9 months) | 28.6 | 40.0 | 50.0
  Other Veg (3 months): number analyzed (Participants) | 8 | 5 | 8
  Other Veg (3 months) | 25.0 | 40.0 | 25.0
  Other Veg (6 months): number analyzed (Participants) | 7 | 5 | 7
  Other Veg (6 months) | 57.2 | 40.0 | 42.9
  Other Veg (9 months): number analyzed (Participants) | 7 | 5 | 6
  Other Veg (9 months) | 42.9 | 50.0 | 50.0
  Citrus (3 months): number analyzed (Participants) | 8 | 5 | 8
  Citrus (3 months) | 12.5 | 20.0 | 0.0
  Citrus (6 months): number analyzed (Participants) | 7 | 5 | 7
  Citrus (6 months) | 0.0 | 0.0 | 0.0
  Citrus (9 months): number analyzed (Participants) | 7 | 5 | 6
  Citrus (9 months) | 0.0 | 60.0 | 0.0
  Fruit (3 months): number analyzed (Participants) | 8 | 5 | 8
  Fruit (3 months) | 25.0 | 80.0 | 25.0
  Fruit (6 months): number analyzed (Participants) | 7 | 5 | 7
  Fruit (6 months) | 28.6 | 60.0 | 42.9
  Fruit (9 months): number analyzed (Participants) | 7 | 5 | 6
  Fruit (9 months) | 71.5 | 80.0 | 33.3
  Whole Milk (3 months): number analyzed (Participants) | 8 | 5 | 8
  Whole Milk (3 months) | 25.0 | 60.0 | 62.5
  Whole Milk (6 months): number analyzed (Participants) | 7 | 5 | 7
  Whole Milk (6 months) | 42.9 | 20.0 | 57.1
  Whole Milk (9 months): number analyzed (Participants) | 7 | 5 | 6
  Whole Milk (9 months) | 42.9 | 20.0 | 66.7
  Low Fat Milk (3 months): number analyzed (Participants) | 8 | 5 | 8
  Low Fat Milk (3 months) | 67.5 | 60.0 | 50.0
  Low Fat Milk (6 months): number analyzed (Participants) | 7 | 5 | 7
  Low Fat Milk (6 months) | 57.1 | 40.0 | 28.6
  Low Fat Milk (9 months): number analyzed (Participants) | 7 | 5 | 6
  Low Fat Milk (9 months) | 42.9 | 40.0 | 16.7
  Eggs (3 months): number analyzed (Participants) | 8 | 5 | 8
  Eggs (3 months) | 12.5 | 0.0 | 25.0
  Eggs (6 months): number analyzed (Participants) | 7 | 5 | 7
  Eggs (6 months) | 14.3 | 0.0 | 28.6
  Eggs (9 months): number analyzed (Participants) | 7 | 5 | 6
  Eggs (9 months) | 28.6 | 20.0 | 16.7
  Whole Grain (3 months): number analyzed (Participants) | 8 | 5 | 8
  Whole Grain (3 months) | 37.5 | 40.0 | 37.5
  Whole Grain (6 months): number analyzed (Participants) | 7 | 5 | 7
  Whole Grain (6 months) | 57.2 | 60.0 | 71.4
  Whole Grain (9 months): number analyzed (Participants) | 7 | 5 | 6
  Whole Grain (9 months) | 57.1 | 60.0 | 50.0
  Pasta (3 months): number analyzed (Participants) | 8 | 5 | 8
  Pasta (3 months) | 12.5 | 20.0 | 12.5
  Pasta (6 months): number analyzed (Participants) | 7 | 5 | 7
  Pasta (6 months) | 0.0 | 20.0 | 14.3
  Pasta (9 months): number analyzed (Participants) | 7 | 5 | 6
  Pasta (9 months) | 14.3 | 0.0 | 16.7
  Baked Goods (3 months): number analyzed (Participants) | 8 | 5 | 8
  Baked Goods (3 months) | 0.0 | 0.0 | 25.0
  Baked Goods (6 months): number analyzed (Participants) | 7 | 5 | 7
  Baked Goods (6 months) | 0.0 | 0.0 | 42.9
  Baked Goods (9 months): number analyzed (Participants) | 7 | 5 | 6
  Baked Goods (9 months) | 0.0 | 0.0 | 33.3
  Beef (3 months): number analyzed (Participants) | 8 | 5 | 8
  Beef (3 months) | 12.5 | 20.0 | 0
  Beef (6 months): number analyzed (Participants) | 7 | 5 | 7
  Beef (6 months) | 28.6 | 20.0 | 14.3
  Beef (9 months): number analyzed (Participants) | 7 | 5 | 6
  Beef (9 months) | 28.6 | 0 | 16.7
  Processed Meat (3 months): number analyzed (Participants) | 8 | 5 | 8
  Processed Meat (3 months) | 0.0 | 0.0 | 0.0
  Processed Meat (6 months): number analyzed (Participants) | 7 | 5 | 7
  Processed Meat (6 months) | 0.0 | 0.0 | 0.0
  Processed Meat (9 months): number analyzed (Participants) | 7 | 5 | 6
  Processed Meat (9 months) | 0.0 | 0.0 | 0.0
  Deep Fried Food (3 months): number analyzed (Participants) | 8 | 5 | 8
  Deep Fried Food (3 months) | 0.0 | 0.0 | 0.0
  Deep Fried Food (6 months): number analyzed (Participants) | 7 | 5 | 7
  Deep Fried Food (6 months) | 0.0 | 0.0 | 0.0
  Deep Fried Food (9 months): number analyzed (Participants) | 7 | 5 | 6
  Deep Fried Food (9 months) | 0.0 | 0.0 | 0.0
  Canned Tuna (3 months): number analyzed (Participants) | 8 | 5 | 8
  Canned Tuna (3 months) | 0.0 | 20.0 | 0.0
  Canned Tuna (6 months): number analyzed (Participants) | 7 | 5 | 7
  Canned Tuna (6 months) | 0.0 | 0.0 | 0.0
  Canned Tuna (9 months): number analyzed (Participants) | 7 | 5 | 6
  Canned Tuna (9 months) | 0.0 | 0.0 | 0.0
  Dark Fish (3 months): number analyzed (Participants) | 8 | 5 | 8
  Dark Fish (3 months) | 0.0 | 0.0 | 0.0
  Dark Fish (6 months): number analyzed (Participants) | 7 | 5 | 7
  Dark Fish (6 months) | 0.0 | 0.0 | 0.0
  Dark Fish (9 months): number analyzed (Participants) | 7 | 5 | 6
  Dark Fish (9 months) | 0.0 | 0.0 | 0.0
  Other Fish (3 months): number analyzed (Participants) | 8 | 5 | 8
  Other Fish (3 months) | 0.0 | 0.0 | 0.0
  Other Fish (6 months): number analyzed (Participants) | 7 | 5 | 7
  Other Fish (6 months) | 0.0 | 0.0 | 0.0
  Other Fish (9 months): number analyzed (Participants) | 7 | 5 | 6
  Other Fish (9 months) | 0.0 | 0.0 | 0.0
  Chicken/Turkey (3 months): number analyzed (Participants) | 8 | 5 | 8
  Chicken/Turkey (3 months) | 12.5 | 0.0 | 25.0
  Chicken/Turkey (6 months): number analyzed (Participants) | 7 | 5 | 7
  Chicken/Turkey (6 months) | 16.7 | 40.0 | 28.6
  Chicken/Turkey (9 months): number analyzed (Participants) | 7 | 5 | 6
  Chicken/Turkey (9 months) | 28.6 | 20.0 | 33.3
  Other Seafood (3 months): number analyzed (Participants) | 8 | 5 | 8
  Other Seafood (3 months) | 0.0 | 20.0 | 0.0
  Other Seafood (6 months): number analyzed (Participants) | 7 | 5 | 7
  Other Seafood (6 months) | 0.0 | 0.0 | 0.0
  Other Seafood (9 months): number analyzed (Participants) | 7 | 5 | 6
  Other Seafood (9 months) | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Exercise Frequency in Women With Gestational Diabetes Post-Partum
Description: This table below shows the average hours per week spent on each activity.
Time Frame: 3 months, 6 months, 9 months, all reported
Population: The "Overall Number of Participants Analyzed" defines the number of participants enrolled in the study.
  The Number in the Rows indicates the number of participants that completed the follow-up surveys required for participation in the study.
  The standard deviation represents the SD from the scores on the scale utilized, not the average numbers per week spent on each activity.
Measure: Mean (Standard Deviation); unit: average hours per week
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
Number analyzed (Participants) | 10 | 8 | 12
average hours per week
  Walking (3 months): number analyzed (Participants) | 8 | 5 | 8
  Walking (3 months) | 3.4 (2.8) | 1.7 (2.35) | 2.2 (1.85)
  Walking (6 months): number analyzed (Participants) | 7 | 5 | 7
  Walking (6 months) | 3.0 (2.99) | 2.2 (2.74) | 2.6 (2.24)
  Walking (9 months): number analyzed (Participants) | 7 | 5 | 6
  Walking (9 months) | 1.6 (2.94) | 0.9 (1.00) | 3.5 (2.43)
  Jogging (3 months): number analyzed (Participants) | 8 | 5 | 8
  Jogging (3 months) | 0 (0.00) | 0.1 (1.30) | 0.1 (1.19)
  Jogging (6 months): number analyzed (Participants) | 7 | 5 | 7
  Jogging (6 months) | 0.2 (1.73) | 0.2 (1.30) | 0.03 (0.76)
  Jogging (9 months): number analyzed (Participants) | 7 | 5 | 6
  Jogging (9 months) | 0.1 (1.13) | 0.3 (1.67) | 0.1 (1.22)
  Running (3 month): number analyzed (Participants) | 8 | 5 | 8
  Running (3 month) | 0 (0.00) | 0.01 (0.45) | 0.1 (1.06)
  Running (6 month): number analyzed (Participants) | 7 | 5 | 7
  Running (6 month) | 0.1 (1.13) | 0.01 (0.55) | 0.03 (0.79)
  Running (9 month): number analyzed (Participants) | 7 | 5 | 6
  Running (9 month) | 0.1 (1.46) | 0.04 (0.89) | 0.1 (1.22)
  Bicycling (3 months): number analyzed (Participants) | 8 | 5 | 8
  Bicycling (3 months) | 0.1 (1.41) | 0.0 (0.00) | 0.0 (0.00)
  Bicycling (6 months): number analyzed (Participants) | 7 | 5 | 7
  Bicycling (6 months) | 0.2 (1.89) | 0.1 (1.34) | 0.1 (1.13)
  Bicycling (9 months): number analyzed (Participants) | 7 | 5 | 6
  Bicycling (9 months) | 0.4 (2.27) | 0.3 (2.24) | 0.0 (0.00)
  Other Aerobic (3 month): number analyzed (Participants) | 8 | 5 | 8
  Other Aerobic (3 month) | 0.0 (0.12) | 0.0 (0.00) | 0.0 (0.00)
  Other Aerobic (6 month): number analyzed (Participants) | 7 | 5 | 7
  Other Aerobic (6 month) | 0.3 (0.60) | 0.03 (0.30) | 0.02 (0.25)
  Other Aerobic (9 month): number analyzed (Participants) | 7 | 5 | 6
  Other Aerobic (9 month) | 0.1 (0.50) | 1.2 (1.88) | 0.4 (0.66)
  Yoga/Stretching (3 months): number analyzed (Participants) | 8 | 5 | 8
  Yoga/Stretching (3 months) | 0.3 (2.14) | 0.3 (1.73) | 0.5 (1.89)
  Yoga/Stretching (6 months): number analyzed (Participants) | 7 | 5 | 7
  Yoga/Stretching (6 months) | 0.1 (1.29) | 1.04 (2.92) | 0.3 (1.99)
  Yoga/Stretching (9 months): number analyzed (Participants) | 7 | 5 | 6
  Yoga/Stretching (9 months) | 0.1 (1.13) | 0.6 (2.68) | 0.4 (1.67)
  Other Vigorous Activity (3 months): number analyzed (Participants) | 8 | 5 | 8
  Other Vigorous Activity (3 months) | 0.5 (2.31) | 0.3 (2.12) | 0.4 (1.93)
  Other Vigorous Activity (6 months): number analyzed (Participants) | 7 | 5 | 7
  Other Vigorous Activity (6 months) | 0.2 (2.04) | 0.9 (2.77) | 0.4 (2.24)
  Other Vigorous Activity (9 months): number analyzed (Participants) | 7 | 5 | 6
  Other Vigorous Activity (9 months) | 0.9 (2.75) | 0.7 (2.00) | 0.5 (2.07)
  Arm Weights (3 months): number analyzed (Participants) | 8 | 5 | 8
  Arm Weights (3 months) | 0.1 (1.41) | 0.2 (1.73) | 0.1 (1.19)
  Arm Weights (6 months): number analyzed (Participants) | 7 | 5 | 7
  Arm Weights (6 months) | 0.2 (1.91) | 0.5 (2.35) | 0.1 (1.25)
  Arm Weights (9 months): number analyzed (Participants) | 7 | 5 | 6
  Arm Weights (9 months) | 0.2 (1.57) | 0.7 (2.83) | 0.2 (1.37)
  Leg Weights (3 months): number analyzed (Participants) | 8 | 5 | 8
  Leg Weights (3 months) | 0.004 (0.35) | 0 (0.00) | 0.04 (0.93)
  Leg Weights (6 months): number analyzed (Participants) | 7 | 5 | 7
  Leg Weights (6 months) | 0.02 (0.76) | 0.5 (2.49) | 0.1 (1.25)
  Leg Weights (9 months): number analyzed (Participants) | 7 | 5 | 6
  Leg Weights (9 months) | 0.0 (0.00) | 0.7 (2.83) | 0.3 (1.76)
  Standing Total (3 months): number analyzed (Participants) | 8 | 5 | 8
  Standing Total (3 months) | 15.9 (1.30) | 8.8 (1.00) | 21.0 (1.51)
  Standing Total (6 months): number analyzed (Participants) | 7 | 5 | 7
  Standing Total (6 months) | 20.8 (1.63) | 10.6 (1.58) | 10.5 (1.17)
  Standing Total (9 months): number analyzed (Participants) | 7 | 5 | 6
  Standing Total (9 months) | 22.7 (2.29) | 19.2 (2.07) | 24.7 (1.22)
  Standing At Home (3 months): number analyzed (Participants) | 8 | 5 | 8
  Standing At Home (3 months) | 13.5 (1.06) | 16.2 (1.00) | 19.9 (1.25)
  Standing At Home (6 months): number analyzed (Participants) | 7 | 5 | 7
  Standing At Home (6 months) | 21.4 (1.46) | 11.9 (1.14) | 11.8 (0.98)
  Standing at Home (9 months): number analyzed (Participants) | 7 | 5 | 6
  Standing at Home (9 months) | 24.4 (2.56) | 9.1 (1.00) | 8.9 (1.47)
  Sitting Total (3 months): number analyzed (Participants) | 8 | 5 | 8
  Sitting Total (3 months) | 17.3 (1.91) | 10.0 (2.08) | 17.4 (1.49)
  Sitting Total (6 months): number analyzed (Participants) | 7 | 5 | 7
  Sitting Total (6 months) | 20.5 (1.35) | 20.0 (1.92) | 28.5 (1.81)
  Sitting Total (9 months): number analyzed (Participants) | 7 | 5 | 6
  Sitting Total (9 months) | 18.4 (1.21) | 18.4 (1.95) | 33.6 (2.43)
  Sitting to Watch TV (3 months): number analyzed (Participants) | 8 | 5 | 8
  Sitting to Watch TV (3 months) | 6.9 (1.58) | 4.8 (0.58) | 13.3 (1.51)
  Sitting to Watch TV (6 months): number analyzed (Participants) | 7 | 5 | 7
  Sitting to Watch TV (6 months) | 6.2 (0.84) | 5.5 (1.58) | 8.6 (1.38)
  Sitting to Watch TV (9 months): number analyzed (Participants) | 7 | 5 | 6
  Sitting to Watch TV (9 months) | 5.0 (1.57) | 6.8 (1.52) | 8.4 (1.17)
  Other Sitting (3 months): number analyzed (Participants) | 8 | 5 | 8
  Other Sitting (3 months) | 11.5 (1.28) | 6.2 (0.58) | 10.0 (0.71)
  Other Sitting (6 months): number analyzed (Participants) | 7 | 5 | 7
  Other Sitting (6 months) | 6.6 (1.13) | 7.5 (0.84) | 6.9 (0.76)
  Other Sitting (9 months): number analyzed (Participants) | 7 | 5 | 6
  Other Sitting (9 months) | 3.4 (1.11) | 4.3 (0.45) | 6.4 (1.05)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events were reported or documented for this study, as it was an education-intervention study that only required survey answers over the course of 1 year (3 month, 6 month, 9 month, 1 year).
Arm/Group | Standard Care | Standard Care+Education Classes | Standard Care+Education Classes+Glucose Monitoring
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/12

LIMITATIONS AND CAVEATS:
Difficulty enrolling and retaining patients for the study; high survey completion but lack of online intervention education modules completion; lack of patient follow up with primary care provider for weights and glucose 1yr postpartum; pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT01681147/Prot_SAP_000.pdf
  • Informed Consent Form (2014-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT01681147/ICF_001.pdf